CLINICAL TRIAL: NCT02795741
Title: Pilot Study to Evaluate the Effects of the Nanohealth, Inc. Cooling Bolero in Women With Common Menopause Symptoms
Brief Title: Study to Evaluate the Effects of the Cooling Bolero in Women With Common Menopause Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Collaborators: Nanohealth, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-16-661
Record Dates: First submitted 2016-06-02; First posted 2016-06-10 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Menopause Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cooling Bolero (Experimental): All participants will use the Cooling Bolero for one month
  Interventions: Device: Cooling Bolero

INTERVENTIONS:
Device: Cooling Bolero — a vest filled with a new material (not ice or a gel) that provides controlled cooling by absorbing heat

SUMMARY:
The Cooling Bolero is a a vest filled with a new material (not ice or a gel) that provides controlled cooling by absorbing heat. The vest is manufactured by Nanohealth. It intended to provide moderate cooling (~15C/59F) through indirect contact with the skin. The material in the device is safe, non-toxic, and eco-friendly.

Recent anecdotal studies of women with common peri-menopausal and menopausal symptoms (hot flashes, night sweats, flushing/sweating of face and neck, and intermittent sleep disturbances) have shown a reduction in both the frequency and intensity of those symptoms after using the Cooling Bolero. Specific (moderate) temperature cooling of the neck and upper torso appears to target and mitigate these common menopausal symptoms. This pilot study attempts to collect additional data on the effects of the Cooling Bolero.

DETAILED DESCRIPTION:
Participants who have consented for this study will first be asked to complete a Baseline Assessment of their menopausal symptoms, including documentation of their baseline weight. If the assessment indicates that the participant has at least 'moderate' menopausal symptoms, then she will then enter the Run-In Period.

During the two-week Run-In Period, participants will use a Symptom Diary for to document the frequency and severity of their menopausal symptoms. At the start of Week 3, participants will return their completed Run-In Period Symptom Diary and receive their Cooling Bolero with instructions on how to use the product during the Treatment Period.

During the Treatment Period, participants should use the Cooling Bolero at least two times per day (morning and evening) for one hour. As feasible, the participant should start to wear the product 30 minutes prior to meal time for these two applications. The participant may also wear the product at additional times, as desired. All applications of the Cooling Bolero during the four-week Treatment Period are to be documented in the Product/Symptom Diary. During the Treatment Period, the participant will also continue to document the frequency and severity of their menopausal symptoms in the Product/Symptom Diary.

At the end of Week 6, the participant will stop using the Cooling Bolero. She will be asked to complete a Product Assessment and have her weight documented.

Participants will be contacted at Week 10 to ask about the status of menopausal symptoms after four weeks of not using the Cooling Bolero.

ELIGIBILITY:
Inclusion Criteria:

* Female, who is at least 18 years old.
* Self-reports having at least two (2) daily hot flashes associated with menopause.

Exclusion Criteria:

• Has another existing medical condition that would prevent study compliance.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07; Primary Completion 2018-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with a reduction in the frequency and/or intensity of menopause symptoms | one month
  Diaries will be used to capture data pre-intervention, during the intervention, and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: David Abramson, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.englewoodhealth.org